CLINICAL TRIAL: NCT01183156
Title: Re-invitation to Screening Colonoscopy: a Randomized Controlled Trial of Reminding Letter and Educational Intervention on Attendance in Nonresponders to Initial Invitation to Screening Colonoscopy
Brief Title: Re-invitation to Screening Colonoscopy: a Randomized Study
Acronym: REINVITE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Malgorzata Pisera, Maria Sklodowska-Curie Memorial Cancer Center, Institute of Oncology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NR13002404
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Colorectal Cancer; Screening; Patient Participation
Keywords: Colorectal Cancer; Screening; Colonoscopy; Attendance; Participation
MeSH Terms: conditions — Colorectal Neoplasms; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Re-invitation letter (Active Comparator)
  Interventions: Behavioral: Re-invitation letter
- Educational Meeting (Active Comparator)
  Interventions: Behavioral: Invitation to educational meeting

INTERVENTIONS:
Behavioral: Re-invitation letter — Re-invitation letter sent 6 weeks prior to prespecified screening colonoscopy appointment date and followed by reminder letter within 3 weeks if no response is received.
  Arms: Re-invitation letter
Behavioral: Invitation to educational meeting — Invitation will be sent 6 weeks prior to educational meeting date and followed by a reminding letter 3 weeks later. Educational meetings will be held in a local culture developement centers and conducted by a medical team responsible for the Polish Colorectal Cancer Screening Program. The aim of the meeting is to overcome barriers to screening colonoscopy. The program of the meeting is tailored to individual needs, doubts, and concerns of the participating group as assessed using brief survey at the beginning of the meeting. The major points to be discussed are: risk and benefit of screening, colorectal cancer risk, pain and sedation, preparation to colonoscopy, consecutive stages of the procedure, comfort and embarrassment.
  Arms: Educational Meeting

SUMMARY:
The aim of this study is to compare the effect of reminding letter and educational intervention on attendance to screening colonoscopy in nonresponders to initial invitation to screening colonoscopy.

DETAILED DESCRIPTION:
NordICC (The NordICC Initiative on Colorectal Cancer, NCT00883792) is a multicenter randomised trial to investigate the effect of screening colonoscopy on CRC incidence and mortality. In Poland, in Warsaw area, at least 10,000 subjects 55-64 years of age are to be invited to screening colonoscopy. A personal letter of invitation containing date and hour of appointment is mailed to every individual randomised to the screening group. Up to 60% of invitees do not respond to the initial invitation and reminding letter. The aim of this study is to compare the effect of reminding letter and educational intervention on attendance to screening colonoscopy in nonresponders to initial invitation to screening colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 55-64 years of age invited for screening colonoscopy within the NordICC trial (NCT00883792) in Poland, who have not responded to the first invitation.

Exclusion Criteria:

* Resident abroad
* Return of unopened letter of invitation and/or reminder (address unknown)
* Message from neighbour/family/post office on death of screenee (not updated in Population Registry).

Ages: 55 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Attendance to screening colonoscopy | 6 months from the date of re-invitation or invitation to educational meeting
  Percentage of invitees attending screening colonoscopy

SECONDARY OUTCOMES:
Response rate to the re-invitation letter or invitation to the educational meeting | 3 months from the date of reinvitation letter or date of invitation to the educational meeting
  Percentage of invitees sending back reply form

CONTACTS AND LOCATIONS:
Overall Officials: Regula Jaroslaw, MD, PhD, Study Director — Center of Oncology Institute and the Maria Sklodowska-Curie Memorial Cancer Center; Malgorzata Pisera, MSc, Principal Investigator — Center of Oncology Institute and the Maria Sklodowska-Curie Memorial Cancer Center; Michal F Kaminski, MD, Study Chair — Center of Oncology Institute and the Maria Sklodowska-Curie Memorial Cancer Center
Locations (1):
- Maria Sklodowska-Curie Memorial Cancer Center, Institute of Oncology, Warsaw, Poland

REFERENCES:
- [Derived] Pisera M, Kaminski MF, Kraszewska E, Rupinski M, Regula J. Reinvitation to screening colonoscopy: a randomized-controlled trial of reminding letter and invitation to educational meeting on attendance in nonresponders to initial invitation to screening colonoscopy (REINVITE). Eur J Gastroenterol Hepatol. 2016 May;28(5):538-42. doi: 10.1097/MEG.0000000000000578. PMID 26967693